CLINICAL TRIAL: NCT06552858
Title: Fluzoparib Combined With Dalpiciclib for Platinum Resistant Recurrent Ovarian Cancer: a Phase II Clinical Study
Brief Title: Fluzoparib Combined With Dalpiciclib for Platinum Resistant Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Director of Gynecological Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-OCR-2024
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; platinum resistance; Fluzoparib; Dalpiciclib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib; dalpiciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib with Dalpiciclib (Experimental): Oral administration of Fluzoparib with Dalpiciclib until disease progression or toxicity intolerance.
  Interventions: Drug: Fluzoparib; Drug: Dalpiciclib

INTERVENTIONS:
Drug: Fluzoparib — 150mg oral bid. A PARP inhibitor that mainly exerts its inhibitory effect on tumor cells by inhibiting DNA repair.
Drug: Dalpiciclib — 150mg oral qd d1-21, q4w. Inhibitor of Cyclin D-CDK4/6 that can inhibit the cell cycle, thereby inducing cell apoptosis.

SUMMARY:
This study aims to investigate the safety and efficacy of combination therapy of Fluzoparib combined With Dalpiciclib for platinum-resistant recurrent ovarian cancer through a single-center, prospective, single-arm, phase II clinical trial, to improve the overall treatment level and prognosis of platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
1. Overall Design: This trial is a single-center, prospective, single-arm, phase II clinical trial to evaluate the safety and efficacy of combination therapy of Fluzoparib combined With Dalpiciclib for platinum-resistant recurrent ovarian cancer.
2. Experimental observation indicators: 1) Main indicators: progression-free survival (PFS), 2) Other indicators: overall survival (OS), objective response rate (ORR), and adverse reactions.
3. Sample size calculation: The median PFS of platinum-resistant recurrent ovarian cancer patients is 3.8 months. In comparison, the experimental group is expected to have a median PFS of 7 months, with an alpha value of 0.05. Following up for 1 year and considering a 10% dropout rate, this study plans to include 30 platinum-resistant recurrent ovarian cancer patients.
4. Data Processing: Enter data and use SPSS statistical software for statistical analysis. Statistical analyst: Clinical Statistics Department of Fudan University Cancer Hospital. Mailing address: 270 Dong'an Road, Shanghai.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old;
2. Sign the informed consent form;
3. Histologically-confirmed epithelial ovarian or fallopian-tube cancer or primary peritoneal cancer.
4. Tumor recurrence or progression within 6 months after using platinum-based drugs;

Exclusion Criteria:

1. Any uncontrolled medical condition that may put the patient at high risk during treatment .
2. Receipt of any other investigational medicinal product within the last 30 days before randomization.
3. Patients with ovarian cancer excluded by pathological or clinical diagnosis;
4. Physical intolerance patients;
5. Patients who are unwilling to participate in the clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Two years
  Progression free survival

SECONDARY OUTCOMES:
OS | Two years
  Overall Survival
ORR | Two years
  Overall Remission Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university shanghai cancer center, Deparment of gynecologic oncology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No